CLINICAL TRIAL: NCT05260255
Title: The Effect of Vitamin D Supplementation on Disease Activity of Systemic Lupus Erythematosus Patients: a Randomized Clinical Trial in Rajavithi Hospital
Brief Title: Effect of Vitamin D Supplement on Disease Activity in SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64013
Record Dates: First submitted 2021-05-12; First posted 2022-03-02 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2021-05

CONDITIONS: Vitamin D Deficiency; Hypocalcemia; Hyperparathyroidism; Systemic Lupus Erythematosus (Disorder)
Keywords: Hypocalcemia; Hyperparathyroidism; End Stage Renal Disease (ESRD); calcitriol; Systemic Lupus Erythematosus ( SLE )
MeSH Terms: conditions — Vitamin D Deficiency; Hypocalcemia; Hyperparathyroidism; Lupus Erythematosus, Systemic; Kidney Failure, Chronic | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D supplementation (Experimental): add on vitamin D2 ( calciferol ) 40,000 IU/wk for 12 weeks
  Interventions: Drug: vitamin D2 ( calciferol )
- placebo (Placebo Comparator): add on placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vitamin D2 ( calciferol ) — add on vitamin D2( calciferol ) 40,000 IU/wk ( 2 cap) for 12 weeks
  Arms: vitamin D supplementation
Drug: Placebo — add on placebo ( 2 cap ) for 12 weeks
  Arms: placebo

SUMMARY:
To study the effect of vitamin D supplementation on disease activity of SLE ( SLEDAI-2K ) and IL-6 level

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year-old
* SLE classified by revised ACR criteria, SLICC 2012 criteria
* SLE patients who have mild to moderate disease activity ( clinical SLEDAI-2K 3-10 ) and has vitamin D level < 40 ng/ml
* currently treated with stable dose of 1 or more of the following background medication : NSAIDs, anti-malarial, MMF, Azathioprine, methotrexate, cyclosporin for at least 1 month, corticosteroid </= 20 mg/d of prednisolone or equivalent dose for at least 2 weeks
* received calciferol 20,000 IU/wk (1 cap) at least 12 weeks

Exclusion Criteria:

* patients with chronic liver disease, CKD stage 3, bed ridden, malignancy
* patients who received drug that interfere with vitamin D metabolism
* poor drug compliance
* overlap with other connective tissue disease or a diagnosis of MCTD
* hx of vitamin D allergy
* hx on MTV or other supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To examine the effect of vitamin D supplementation on SLE disease activity | 12 weeks
  Study the SLE disease activity by SLEDAI-2K in relation with vitamin D levels

SECONDARY OUTCOMES:
To examine the effect of vitamin D supplementation on IL-6 level | 12 weeks
  monitor serum vitamin D before and after intervention
To determine whether IL-6 can early detection in SLE disease flare | 12 weeks
  monitor serum IL-6 before and after intervention compare with SLE disease activity index ( SLEDAI-2K )
To determine adverse reaction of high dose vitamin D | 12 weeks
  monitor adverse reaction of vitamin D after intervention
To study the effect of vitamin D supplementation on anti-dsDNA titer | 12 weeks
  monitor serum anti-dsDNA titer before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ding J, Su S, You T, Xia T, Lin X, Chen Z, Zhang L. Serum interleukin-6 level is correlated with the disease activity of systemic lupus erythematosus: a meta-analysis. Clinics (Sao Paulo). 2020 Oct 19;75:e1801. doi: 10.6061/clinics/2020/e1801. eCollection 2020. PMID 33084768
- [Background] Hassanalilou T, Khalili L, Ghavamzadeh S, Shokri A, Payahoo L, Bishak YK. Role of vitamin D deficiency in systemic lupus erythematosus incidence and aggravation. Auto Immun Highlights. 2017 Dec 26;9(1):1. doi: 10.1007/s13317-017-0101-x. PMID 29280010
- [Background] Aranow C, Kamen DL, Dall'Era M, Massarotti EM, Mackay MC, Koumpouras F, Coca A, Chatham WW, Clowse ME, Criscione-Schreiber LG, Callahan S, Goldmuntz EA, Keyes-Elstein L, Oswald M, Gregersen PK, Diamond B. Randomized, Double-Blind, Placebo-Controlled Trial of the Effect of Vitamin D3 on the Interferon Signature in Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2015 Jul;67(7):1848-57. doi: 10.1002/art.39108. PMID 25777546